CLINICAL TRIAL: NCT05967117
Title: Chest CT Using Low-concentration Iodine Contrast Media - a Prospective Multicenter Comparative Study
Brief Title: Chest CT Using Low-concentration Iodine Contrast Media
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jung Im Jung (Other)
Collaborators: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jung Im Jung, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CTC42M014
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases | interventions — Iohexol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chest CT evaluation (Administrate contrast media for CECT) (Active Comparator): Patients who are planned chest contrast enhanced CT scan ; Conventional concentration iodine contrast agents with the conventional tube voltage
  Interventions: Drug: Iohexol (320mgI/mL) with 120kVp
- Chest CT evaluation (Experimental 1) (Experimental): Patients who are planned chest contrast enhanced CT scan ; Conventional concentration iodine contrast agents with the low tube voltage
  Interventions: Drug: Iohexol (320mgI/mL) with 100kVp
- Chest CT evaluation (Experimental 2) (Experimental): Patients who are planned chest contrast enhanced CT scan ; Low concentration iodine contrast agents with the low tube voltage)
  Interventions: Drug: Iohexol (270mgI/mL) with 100kVp
- Chest CT evaluation (Experimental 3) (Experimental): Patients who are planned chest contrast enhanced CT scan; Ultra Low concentration iodine contrast agents with the low tube voltage)
  Interventions: Drug: Iohexol (240mgI/mL) with 100kVp

INTERVENTIONS:
Drug: Iohexol (320mgI/mL) with 120kVp — Patient undergoing CT scan with 120kVp protocol and using Iobrix inj. 320 (Taejoon pharm, Seoul, South Korea). CT images were obtained 55sec after Contrast media injection(100mL, 2mL/sec) with 20mL saline flushing.
  Other Names: Iobrix inj. 320
  Arms: Chest CT evaluation (Administrate contrast media for CECT)
Drug: Iohexol (320mgI/mL) with 100kVp — Patient undergoing CT scan with 100kVp protocol and using Iobrix inj. 320 (Taejoon pharm, Seoul, South Korea). CT images were obtained 55sec after Contrast media injection(100mL, 2mL/sec) with 20mL saline flushing.
  Other Names: Iobrix inj. 320
  Arms: Chest CT evaluation (Experimental 1)
Drug: Iohexol (270mgI/mL) with 100kVp — Patient undergoing CT scan with 100kVp protocol and using Iobrix inj. 270 (Taejoon pharm, Seoul, South Korea). CT images were obtained 55sec after Contrast media injection(100mL, 2mL/sec) with 20mL saline flushing.
  Other Names: Iobrix inj. 270
  Arms: Chest CT evaluation (Experimental 2)
Drug: Iohexol (240mgI/mL) with 100kVp — Patient undergoing CT scan with 100kVp protocol and using Iobrix inj. 240 (Taejoon pharm, Seoul, South Korea). CT images were obtained 55sec after Contrast media injection(100mL, 2mL/sec) with 20mL saline flushing.
  Other Names: Iobrix inj. 240
  Arms: Chest CT evaluation (Experimental 3)

SUMMARY:
This study aims to evaluate the quality of images when low-concentration iodine contrast agents is used in chest CT with low tube voltage and if they can be used in routine imaging.

The primary endpoint of the study was the quality of the image and comparison of chest CT by using low and conventional concentration iodine contrast agents with low tube voltage and chest CT by using the conventional concentration iodine contrast agents with the conventional tube voltage; The secondary endpoint is optimizing chest CT protocol using an iodine contrast agent.

DETAILED DESCRIPTION:
With persistent advances in computed tomography (CT) technology, there is a need for continuous investigation and optimization of injection protocols. Intravenous contrast enhancement in CT is affected by various interacting factors, which can be roughly divided into 3 categories: patient, contrast medium and CT scanning. Over the last decade, evolutions in technology has resulted in faster CTs with improved temporal and spatial resolutions; newer techniques such as iterative reconstruction has enabled lower tube voltage (expressed in units of peak kiloVolt, kVp) and lower dose CTs with less noise and preserved image quality. As CT scanning is one of the major determinants of contrast enhancement at CT, such technological advances in CT can be assumed to have invariably caused alterations in the degree of contrast enhancement at CT. However, despite changes in CT scanning techniques, recommended contrast injection protocol for chest CT with enhancement (CECT), including concentration of iodine contrast material, have not changed over the last decade; for routine chest CECT, the use of 300-350 mgI/ml iodine contrast material has been recommended without definitely stating the precise reasons using that specific iodine concentration.

Therefore, the aim of this study was to evaluate the image quality of low voltage chest CECT using LCCM(Low-Concentration Iodinated Contrast Media.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older, weighing less than 90 kg, and BMI less than 30 who underwent contrast-enhanced chest CT alone

Exclusion Criteria:

1. Under the age of 18
2. Cases where contrast-enhanced CT cannot be performed
3. Heart failure
4. Pregnancy
5. If patients cannot voluntarily give written consent to participate in this clinical trial
6. In the case of an anatomical deformation that may interfere with image analysis in the previous image
7. Patients with a history of hypersensitivity to IOBRIX, components of IOBRIX, and iodine-based drugs
8. Patients with severe thyroid disease (Iodine may accumulate in the thyroid gland and worsen symptoms.)
9. Those who are judged unsuitable by the tester for other reasons Patients aged 19 years or older, weighing less than 90 kg, and BMI less than 30 who underwent contrast-enhanced chest CT alone

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Anatomic depiction (including image sharpness) | 12 months after the CT scan (Chest contrast-enhanced CT is a 1-day procedure, but evaluating all the images will be done one year after the 1st CT scan.)
  3 points scale qualitative analysis evaluated by two different radiologists (Poor, moderate, excellent)
Noise | 12 months after the CT scan
  3 points scale qualitative analysis evaluated by two different radiologists (Severe, minor, negligible)
Contrast-related artifact | 12 months after the CT scan
  3 points scale qualitative analysis evaluated by two different radiologists (Severe, minor, negligible)
Overall diagnostic acceptability | 12 months after the CT scan
  5 points scale qualitative analysis evaluated by two different radiologists (Non-diagnostic, suboptimal, standard, better than standard, Excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Im Jung, MD, PhD, Study Chair — Seoul St. Mary's Hospital
Locations (6):
- South Korea (6):
  - Bucheon St. Mary's Hospital, The Catholic University of Korea, Bucheon-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, Seocho-gu
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No